CLINICAL TRIAL: NCT01390610
Title: Observational Evaluation Using Continuous Glucose Monitoring to Determine Timing and Frequency of Self-Monitored Blood Glucose by Therapy Type in Patients With Type 2 Diabetes (REACT-4 Matrix Definition Study)
Brief Title: Continuous Glucose Monitoring Self-Monitored Blood Glucose Type 2 Therapy Matrix Definition
Acronym: REACT4
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: 04111-11-C
Record Dates: First submitted 2011-06-29; First posted 2011-07-11 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Blood Glucose Monitoring
Keywords: Continuous Glucose Monitoring; Self Monitored Blood Glucose; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to use data from the Continuous Glucose Monitoring (CGM) device and your Self-Monitored Blood Glucose (SMBG) levels to determine the best times to test blood glucose levels using SMBG.

DETAILED DESCRIPTION:
The investigators propose to employ CGM technology in subjects using insulin sensitizers, incretin mimetics and potentiators, insulin secretagogues and insulin to identify the minimum episodic data set that closely mimics CGM data. Specifically, the investigators propose to employ blinded CGM for 2 weeks to capture the diurnal glucose patterns of individuals on different therapeutic regimens. The investigators propose to examine these data to determine whether a specific pattern of SMBG testing derived from these data would provide the same information (e.g., detection of hypoglycemia, measures of glycemic exposure, variability and stability) not possible by relying solely on current SMBG testing schedules.

In preparation for this study the investigators developed a matrix using data collected from previous studies. The matrix summarizes the amount of CGM data the investigators currently possess and indicates where the investigators lack sufficient data to produce SMBG testing schedules based on CGM data. It was determined that 6 cases were needed for each therapy group. An underlying question is whether after the investigators fill this matrix the investigators can discover a common testing pattern for SMBG that would provide sufficient information to uncover the myriad perturbations in glucose patterns that characterize type 2 diabetes. To assure that the investigators are collecting adequate monitoring data, the investigators propose to use Ambulatory Glucose Profile (AGP) analysis of blinded CGM data. This novel approach will enable us to answer the question as to the optimum time and number of SMBG tests sufficient to guide clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Diagnosed with type 2 diabetes and treated with diabetes medication(s) as required by the protocol (See Section 3.1)
* Age 18 and older
* Willing to give informed consent
* Motivated and capable of following the protocol and instructions provided by the healthcare professional
* Available for the study on the scheduled visit days
* Have not participated in a prior research trial at IDC that utilized CGM

Exclusion Criteria:

* Under 18 years of age
* Skin abnormalities at the CGM insertion sites that would confound assessment of the effect of the device on the skin
* Allergy to adhesives
* Taken prednisone or cortisone medications in the previous 30 days
* Currently pregnant or planning pregnancy during the study period
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* Unable to follow the study protocol
* Unable to speak, read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty seven persons with type 2 diabetes age 18 and older.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Derive optimum Self Monitored Blood Glucose (SMBG) testing patterns from CGM data. CGM data will be graphically and statistically represented by an Ambulatory Glucose Profile (AGP). | 2 weeks of CGM data

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Mazze, PhD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States